CLINICAL TRIAL: NCT03392389
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1653, a Combined Human Metapneumovirus and Human Parainfluenza Virus Type 3 Vaccine, When Administered to Healthy Adults
Brief Title: Safety, Reactogenicity, and Immunogenicity of mRNA-1653 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: mRNA-1653-P101
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Human Metapneumovirus and Human Parainfluenza Infection
Keywords: mRNA-1653; human metapneumovirus; human parainfluenza vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1653 (Experimental)
  Interventions: Biological: mRNA-1653
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1653 — Escalating dose levels
  Arms: mRNA-1653
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
This clinical study will assess the safety, reactogenicity and immunogenicity of mRNA-1653, a combined human metapneumovirus and human parainfluenza virus type 3 vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to comply with the study procedures and provides written informed consent
* 18 to 49 years of age
* Body mass index between 18 and 35 kg/m2
* In good health based on medical history, physical examination, vital sign measurements and laboratory safety tests performed prior to initial study vaccination
* Negative urine pregnancy test at the screening visit and the day of each vaccination for females of childbearing potential
* Female subjects must either be of non-childbearing potential or use acceptable methods of contraception from at least 30 days prior to enrollment and through 3 months following last vaccination
* Willing to comply with the requirements of the protocol (eg, complete Diary Cards, return for follow-up visits, be available for safety phone calls)

Exclusion Criteria:

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care
* A history of malignancy in the last 10 years
* If female and of childbearing potential, is pregnant or lactating, has not adhered to an adequate contraception method from at least 30 days before study entry, or does not plan to do so for at least 3 months after the last vaccination
* Abnormal screening safety laboratory test results including liver enzyme tests
* Administration of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine or has plans for administration during the study period
* Prior administration of investigational agent using lipid nanoparticle formulations
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies
* A positive test result for drugs of abuse
* Chronic administration of potentially hepatotoxic drugs or have other medical conditions that affect the liver (eg, alcohol abuse)
* A history of idiopathic urticaria
* Plans for administration or has been administered a vaccine within the period from 30 days before through 30 days after each study vaccination, with the exception of any licensed influenza vaccine administered ≥15 days before or after any study vaccination
* Any chronic administration of an immunosuppressant or other immune modifying drug
* Prior administration of immunoglobulins and/or any blood products within the 3 months before the first study vaccine or has plans for administration during the study period
* Any known or suspected immune-mediated disease or immunosuppressive condition as determined by medical history and/or physical examination
* A history of hypersensitivity or serious reactions to previous vaccinations
* Any bleeding disorder considered a contraindication to IM injection or blood draw
* Any acute illness or fever at screening
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject if enrolled or could interfere with evaluation of the study drug or interpretation of study results
* Donation of blood or blood products > 450 mL within 30 days of dosing.
* Is an immediate family member or household member of study personnel

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited AEs (local and systemic reactogenicity events) | 7 days following each dose administration
Frequency of unsolicited adverse events | 28 days following each dose administration
Frequency of serious adverse events (SAE), adverse events of special interest (AESI), and medically-attended AEs | one year following the last dose administration
Frequency of clinical laboratory adverse events | 1 month following the last dose administration
Geometric mean titer (GMT) of the serum anti-hMPV and anti-PIV3 neutralizing antibodies | 1 month following the last dose administration
Proportion of subjects with a ≥ 4-fold increase in serum anti-hMPV and anti-PIV3 neutralizing antibody titer from baseline to post-vaccination | 1 month following the last dose administration
Proportion of subjects who achieve serum anti-hMPV and anti-PIV3 neutralizing antibody titers greater than the third quartile of the serum anti-hMPV and anti-PIV3 antibody titers overall distribution at baseline | 1 month following the last dose administration

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of the serum anti-hMPV and anti-PIV3 neutralizing antibodies | 6 months and 1 year following the last dose administration
Proportion of subjects with a ≥ 4-fold increase in serum anti-hMPV and anti-PIV3 neutralizing antibody titer from baseline to post-vaccination | 6 months and 1 year following the last dose administration
Proportion of subjects who achieve serum anti-hMPV and anti-PIV3 neutralizing antibody titers greater than the third quartile of the serum anti-hMPV and anti-PIV3 antibody titers overall distribution at baseline | 6 months and 1 year following the last dose administration

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Benchmark Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No